CLINICAL TRIAL: NCT07384585
Title: Feasibility of Light Therapy in the Pediatric ICU
Brief Title: Feasibility of Light Therapy in the Pediatric Intensive Care Unit (ICU)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Beth Kalvas (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Laura Beth Kalvas, Nurse Scientist, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005565
Record Dates: First submitted 2026-01-21; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Circadian Dysregulation; Light Exposure; Pediatric Critical Illness
MeSH Terms: conditions — Chronobiology Disorders | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Light Therapy (Experimental)
  Interventions: Other: Light Therapy

INTERVENTIONS:
Other: Light Therapy — Light therapy will be delivered via a light box for a maximum of 5 days in the pediatric ICU. Light therapy will be initiated 1 to 2 hours following participant's typical wake time, and continue for 3 hours. The light box light intensity is 10,000 lux with high blue light content (5,000 Kelvin). The light box blocks ultraviolet rays. The portable light box will be placed in front or to the side of the child at a distance of 2 feet. The light box can be moved with activity and turned off at any time if requested by the child, family, or staff.
  Other Names: bright light exposure

SUMMARY:
The goal of this clinical trial is to understand how easy or difficult it is for critically ill children (4-17 years old) to have light therapy while in the pediatric ICU. Participants will have a light meter at their bedside to measure light levels. Each morning, a light box will be placed at their bedside. Children, family, and staff will be asked to completed feedback surveys regarding the light therapy. Study participation will continue for a maximum of 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Within 48 hours of pediatric ICU admission at study hospital
* Anticipated to remain admitted to the study hospital pediatric ICU for additional 48 hours
* English-speaking parent/legally authorized representative available at the bedside

Exclusion Criteria:

* Patients unable to open their eyes to receive light therapy (Glasgow Coma Scale eye opening score of 1)
* Patients with contraindications to light therapy (e.g., migraines, retinal disease, diseases associated with retinal complications, blindness, bipolar disorder, traumatic brain injury)
* Suspected/identified neglect/abuse, Child Protective Services involvement, or ward of state
* Children receiving palliative/end-of-life care

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of light therapy for children, families, and staff. | Maximum of 5 days of light therapy.
  Feasibility of light therapy assessed via feedback surveys from children, families, and clinical staff.
Duration of light therapy | Maximum of 5 days of light therapy.
  Hours of light therapy received per study day.

SECONDARY OUTCOMES:
Adverse side effects of light therapy. | Maximum of 5 days of light therapy.
  For each day of light therapy, presence of commonly reported side effects of light therapy (e.g., headache, eye strain, nausea, agitation) will be monitored and recorded in a daily monitoring form. Unanticipated problems and reportable adverse side effects will be monitored and recorded in an adverse event form. Presence of side effects will be determined from speaking with the bedside nurse, parent/caregiver, and child, review of the electronic medical record, and child/family/staff feedback surveys.
Light levels | Maximum of 5 days of light therapy.
  Continuous bedside monitoring of light levels in lux via a light meter.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Results of this small clinical trial testing feasibility of light therapy in the pediatric ICU will be shared in aggregate via publication at presentations at the study hospital and conferences.